CLINICAL TRIAL: NCT06307119
Title: The Effectiveness of Model of Human Occupation-Based Intervention on Occupational Participation in Individuals With Premenstrual Syndrome Symptoms
Brief Title: Model of Human Occupation-Based Intervention on Premenstrual Syndrome Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Berkan Torpil, PhD, Associate Professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-01
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Premenstrual Syndrome
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Occupational Therapy and Relaxation Group (Experimental): MOHO Based Intervention and Jacobson's Progressive Muscle Relaxation method
  Interventions: Behavioral: Occupational Therapy and Relaxation Group
- Relaxation Group (Experimental): Jacobson's Progressive Muscle Relaxation method
  Interventions: Behavioral: Relaxation Group
- Control Group (No Intervention): No İntervention

INTERVENTIONS:
Behavioral: Occupational Therapy and Relaxation Group — MOHO Based Intervention
  The client-centered occupational therapy comprises five distinct stages:
  1. Client-Centered Goal Setting:It involves collaboratively establishing goals the client's needs and aspirations.
  2. Creating the Therapy Plan:Comprehensive therapy plan is devised from the findings from OSA and MOHOST results.
  3. Implementing the Interventions:These interventions aimed addressing various personal challenges,financial management,stress management.
  4. Evaluating the Results:It involves adjusting the therapy plan as needed based on the participant's responses and outcomes.
  5. Receiving Feedback
  Jacobson's Progressive Muscle Relaxation
  Starting with the lower extremities,participants sequentially tensed and relaxed muscle groups,moving from distal to proximal regions,encompassing toes,ankles,thighs,buttocks,abdomen,fingers,triceps,shoulders,and face.During all these stages,it was ensured to maintain contraction for 5 seconds and to relax and rest for 10 seconds.
  Arms: Occupational Therapy and Relaxation Group
Behavioral: Relaxation Group — Jacobson's Progressive Muscle Relaxation (JPMR) Participants underwent training in relaxation techniques involving mental visualization and Jacobson's progressive muscle relaxation method with the aid of music. Starting with the lower extremities, participants sequentially tensed and relaxed muscle groups, moving from distal to proximal regions, encompassing toes, ankles, thighs, buttocks, abdomen, fingers, triceps, shoulders, cervical muscles, and face. During all these stages, it was ensured to maintain contraction for 5 seconds and to relax and rest for 10 seconds.
  Arms: Relaxation Group

SUMMARY:
This study was conducted to examine the effect of two different occupational therapy interventions on premenstrual syndrome symptoms in university students. This study was designed according to the CONSORT statement, which provides a standard method for randomised controlled trial (RCT) design. The study was approved by the Local Ethics Committee. Written informed consent was obtained from all participants before the study.

DETAILED DESCRIPTION:
The current study constituted a single-center, two-arm, parallel-group randomized controlled trial involving university students from a public university in Turkey. Prior to study, the research protocol received approval from the local ethics committee. All participants provided written informed consent. The current study was designed according to the CONSORT statement, which provides a standardized method for randomized controlled trial (RCT) design.

Participants The study employed a convenience sampling method. Invitation messages were sent via WhatsApp to 2500 undergraduate students within the university's Faculty of Health Sciences, where the study was conducted. A total of 230 participants were enrolled in the study and assessed by a researcher (B.T.). According to the inclusion and exclusion criteria, 125 people were excluded. 105 students were divided into three groups: Control Group, Relaxation Group, and Occupational Therapy and Relaxation Group. During the study, 10 participants-3 from group Occupational Therapy and Relaxation Group and 7 from the Relaxation Group -were unable to complete the intervention program. Consequently, the study was concluded with 95 university students with premenstrual syndrome .

Demographic data were gathered prior to randomization. Participants were randomly assigned (allocation ratio of 1:1) to either the Control Group, Relaxation Group, and Occupational Therapy and Relaxation Group. using computer-generated randomization. All participants underwent a 6-week intervention before and after evaluation, which was conducted by the same researcher who was blinded to the group allocation. No monetary or credit compensation was provided for participation in the study.

The data underwent analysis using the SPSS version 26.0 statistical software package. Normality assessment was conducted using the Shapiro-Wilk test. Group differences were assessed using the chi-square test for nominal data and the Mann-Whitney U test for ordinal data. To compare pre- and post-intervention results within groups, the Wilcoxon signed-rank test was employed. Participants who didn't complete the post-evaluation (n = 10) were excluded. Quade's rank analysis of covariance test was utilized to control baseline disparities in measurements. Effect size was calculated to quantify intervention effectiveness relative to comparisons, utilizing means, standard deviations, and correlation coefficients for within-group changes. Effect size benchmarks of 0.20, 0.50, and 0.80 standard deviations were considered small, medium, and large, respectively, according to Cohen (1992). Statistical significance was defined as p < .05.

ELIGIBILITY:
Inclusion Criteria:

* (1) diagnosed with Premenstrual Syndrome as per the Premenstrual Symptom Screening Tool (PSST)
* (2) aged 18 years or older
* (3) maintaining a regular menstrual cycle

Exclusion Criteria:

* (1) diagnosed with another psychiatric or gynecological disorder
* (2) pregnant or breastfeeding
* (3) taking oral contraceptive pills
* (4) receiving hormonal treatment to regulate menstrual cycle
* (5) unable to consistently engage in the intervention program

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-02 (Actual)

PRIMARY OUTCOMES:
Occupational Self-Assessment | 20 minutes
  The Occupational Self-Assessment(OSA) version-2.2 is tool comprising 21 items,aimed at evaluating both occupational competence and value.Each item within the OSA is rated using two distinct 4-point scales.The first scale measures occupational competence,ranging from 1(indicating significant difficulty) to 4(indicating excellent performance).Conversely,the second scale evaluates value,ranging from 1(indicating low importance) to 4(indicating utmost importance).Subsequently,individual item scores are aggregated to derive total scores for both competence and value,which are then standardized to a scale of 0 to 100 following prescribed guidelines.Higher total scores signify elevated levels of both occupational competence and value.Upon completion of the assessment,participants are prompted by the therapist to identify the four items they consider to be of utmost priority.Turkish version of this instrument underwent validation in a prior study conducted by Pekçetin et al. in 2018.

SECONDARY OUTCOMES:
The Model of Human Occupation Screening Tool (MOHOST) | 30 minutes
  The MOHOST,serves as assessment tool aimed at gauging occupational participation,irrespective of specific diagnoses.MOHOST is structured to measure pertinent concepts derived from the Model of Human Occupation(MOHO).Within this framework,each of the six key concept-denoted as (a)volition or motivation for occupations,(b)habituation or patterns of occupation,(c)communication and interaction skills,(d)process skills,(e)motor skills,and (f)environment-is represented by four distinct items.In the MOHOST each of the 24 items is assessed using a four-point rating scale,focusing on its impact on occupational participation.The ratings are as follows:"F" signifies that the item"Facilitates" occupational participation,"A" indicates that the item "Allows" participation,"I" suggests that it "Inhibits" participation,and "R" denotes that the item"Restricts" participation.Low scores on the MOHOST indicate that occupational participation is restricted.Turkish version of MOHOST developed by Zakarneh.

OTHER OUTCOMES:
Premenstrual Symptom Screening Tool | 10 minutes
  We utilized an instrument developed by Ozdel et al. (2015) to assess premenstrual syndrome (PMS) to DSM-V criteria. This scale comprises 25 items that evaluate symptoms associated with PMS. A unified score is derived from the scale, where symptoms are categorized into three subgroups: Premenstrual Dysphoric Disorder (PMDD), PMS, and normal/non-PMDD. The scale demonstrated a Cronbach's alpha coefficient of 0.928, indicating high internal consistency.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Turkey, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No